CLINICAL TRIAL: NCT05337592
Title: A Randomised, Single-blind, Placebo-controlled Trial to Investigate Safety, Tolerability, and Pharmacokinetics of Single Rising Doses of BI 1815368 Administered as Oral Solution to Healthy Male Subjects (SRD Part), and a Randomised, Open-label, Single-dose, Three-way Cross-over Part Investigating Relative Bioavailability of BI 1815368 as Tablet Versus Oral Solution and Tablet With and Without Food in Healthy Male Subjects (BA Part)
Brief Title: A Study in Healthy Men to Test How Different Doses of BI 1815368 Are Tolerated and How BI 1815368 is Taken up in the Body With or Without Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 1485-0001; 2021-006856-16 (EudraCT Number)
Record Dates: First submitted 2022-04-14; First posted 2022-04-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: This study has 2 parts: a single rising dose (SRD) part and a bioavailability (BA) part. For the SRD part the intervention study model is sequential, while for the BA part the intervention study model is crossover.
Who Masked: Participant
Masking Description: For the Single Rising Dose (SRD) part the participant is blinded. For the bioavailability (BA) part no masking is applicable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- SRD part: BI 1815368 (Experimental)
  Interventions: Drug: BI 1815368 formulation 1
- SRD part: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- BA part: T1-R-T2 (Experimental): R: BI 1815368 formulation 1, fasted condition T1: BI 1815368 formulation 2, fasted condition T2: BI 1815368 formulation 2, fed condition
  Interventions: Drug: BI 1815368 formulation 1; Drug: BI 1815368 formulation 2
- BA part: R-T2-T1 (Experimental)
  Interventions: Drug: BI 1815368 formulation 1; Drug: BI 1815368 formulation 2
- BA part: T2-T1-R (Experimental)
  Interventions: Drug: BI 1815368 formulation 1; Drug: BI 1815368 formulation 2

INTERVENTIONS:
Drug: BI 1815368 formulation 1 — BI 1815368 formulation 1
  Arms: BA part: R-T2-T1; BA part: T1-R-T2; BA part: T2-T1-R; SRD part: BI 1815368
Drug: Placebo — Placebo
  Arms: SRD part: Placebo
Drug: BI 1815368 formulation 2 — BI 1815368 formulation 2
  Arms: BA part: R-T2-T1; BA part: T1-R-T2; BA part: T2-T1-R

SUMMARY:
Single-rising dose (SRD) part The main objectives of the SRD part of this trial are to investigate safety, tolerability and pharmacokinetics (PK) of BI 1815368 in healthy male subjects following oral administration of single rising doses.

Bioavailability (BA) part The main objective of the BA part is to investigate the relative bioavailability of a tablet formulation versus oral solution and to assess the influence of food on the relative bioavailability of the tablet formulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP),pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 45 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent in accordance with International Council for Harmonisation- Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Further exclusion criteria apply

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-18 (Actual)

PRIMARY OUTCOMES:
SRD part: Occurrence of any treatment-emergent adverse event | Up to Day 14
BA part: Area under the concentration-time curve of BI 1815368 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | Up to Day 5
BA part: Maximum measured concentration of BI 1815368 in plasma (Cmax) | Up to Day 5

SECONDARY OUTCOMES:
SRD part: Area under the concentration-time curve of BI 1815368 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | up to Day 6
SRD part: Maximum measured concentration of BI 1815368 in plasma (Cmax) | up to Day 6
BA part: Area under the concentration-time curve of BI 1815368 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to Day 5

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com